CLINICAL TRIAL: NCT04234503
Title: Ethical Activity Profile of Nurse Managers -Testing Ethics Quarter as an Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Laura Laukkanen, Principal Investigator, University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EQ-i
Record Dates: First submitted 2020-01-13; First posted 2020-01-21 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Ethics
Keywords: nurse managers; ethical activity profile

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ethics Quarter (Experimental): Nurse managers perform 12 educational packages in web-page www.etiikanvartti.fi.
  Interventions: Behavioral: Ethics Quarter
- Standard organisational ethics structures (No Intervention): Nurse managers continue in their standard organisational ethics structures

INTERVENTIONS:
Behavioral: Ethics Quarter — In the intervention, nurse managers have two educational packages per week, one taking 15 minutes (one quarter).The structure of the whole intervention is made according to the dimensions of ethical activity profile of nurse managers (Laukkanen et al. a2016; Laukkanen et al b2016) consisting of managers:
  1. Developing of own ethics knowledge,
  2. Influencing ethical issues,
  3. Conducting/implementing ethics research,
  4. Identifying and
  5. Solving ethical problems.
  Intervention includes also orientation and summary, in total 12 educational packages.
  After every dimension, NMs have to make self-reflection and development plans, in total five times. This provides them the opportunity to link their everyday experience with ethical theory.
  Arms: Ethics Quarter

SUMMARY:
The aim of this study is:

1. to test a new ethics educational intervention for nurse mangers, Ethics Quarter (EQ) and
2. to measure the feasibility and the usability of the EQ

The detailed research questions and hypothesis of this study are as follows:

1. Is EQ effective in increasing NMs' ethics knowledge?
2. Is EQ effective in increasing NMs' influencing ethics issues?
3. Is EQ effective in increasing NMs' ethics research implementing?
4. Is EQ effective in increasing NMs' ethics problem identifying?
5. Is EQ effective in increasing NMs' ethics problem solving?

   H 1-5: It is hypothesized that participating into EQ promotes NM's ethics knowledge, influencing ethics issues, ethics research implementing, ethics problem identifying and ethics problem solving compared to comparisons.
6. What are NM's perceptions of feasibility and usability of the EQ?

The ultimate goal is to strengthen nurse managers' ethical activity profile and create a new, modern way to promote ethical management of nursing.

DETAILED DESCRIPTION:
A new educational intervention, EQ, for nurse managers has developed. Intervention development has evaluated by using criteria for complex interventions in health care (CReDECI)- guideline (Möhler et al. 2012). EQ intervention is based on distance learning method and it consists of 12 educational packages included in the virtual learning environment www.etiikanvartti.fi.

Effectiveness of EQ intervention will be tested by using an individually randomized controlled trial with baseline-, post- and follow-up-measurements.The intervention group will participate in the educational EQ intervention and the control group will not participate.

Data will be collected via the membership register of the Union of Health and Social Care Professionals in Finland (Tehy) trade union. This union is a national interest group for nurses, nurse managers and advanced consultants/specialists in the social and health-care sector having a Master's degree (nursing science or related) or registered nurses degree.

Based on statistical power analysis, the required sample size for the study will be 87 NMs at both groups, at 80%, 0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* Working as a nurse manager
* Finnish-speaking

Exclusion Criteria:

* Unwilling to provide consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Changes in nurse managers' ethical activity profile level. | Baseline, week 6 and week 10
  Ethical activity profile consists of five dimensions: 1) Developing of own ethics knowledge, 2) Influencing ethical issues, 3) Conducting/implementing ethics research, 4) Identifying and 5) Solving ethical problems.
  Dimensions 1-3 will be measured with Developing, Influencing and implementing ethics -instrument (DIIEI), Dimension 4 will be measured with Ethical Sensitivity Scale Questionnaire (ESSQ) and Dimension 5 will be measured with Nurses' Moral Courage Scale (NMCS) at baseline (before the intervention), week 6 (after the intervention) and week 10.
  Results of the all three instruments create one primary outcome measure, ethical activity profile level. All the instruments are 5-point Likert-scales (1=totally disagree; 5=totally agree/1= Does not describe me at all; 5= Describes me very well) and the higher scores indicate higher self-assessed ethical activity profile level.
Changes in nurse managers' ethical activity profile level. | Baseline, week 6 and week 10
  Changes in nurse managers' self-assessed level of the ethical activity profile measured with the Ethical activity-instrument (EAI) at baseline (before the intervention), week 6 (after the intervention) and week 10. The higher scores indicate higher self-assessed ethical activity profile level.

SECONDARY OUTCOMES:
Changes in nurse managers' knowledge level. | Baseline, week 6 and week 10
  Changes in knowledge level is measured with the Nursing Management Ethics Knowledge-test (NMEKT) at baseline (before the intervention), week 6 (after the intervention) and week 10. The higher scores indicate higher level of knowledge.
Nurse managers' perceptions of the feasibility and usability of EthicsQuarter. | Week 6
  Perceptions of the feasibility is measured with open questions and the usability of the web site is measured with the System Usability Scale (SUS) at week 6. The higher scores indicate higher usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Finland, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laukkanen L, Suhonen R, Poikkeus T, Loyttyniemi E, Leino-Kilpi H. The effectiveness of the Ethics Quarter intervention on the ethical activity profile of nurse managers: A randomized controlled trial. J Nurs Manag. 2022 Oct;30(7):2126-2137. doi: 10.1111/jonm.13411. Epub 2021 Jul 21. PMID 34231275
- See also: Ethical activity profile of nurse managers. — https://doi-org.ezproxy.utu.fi/10.1111/jonm.12348
- See also: Solving work-related ethical problems. — https://doi-org.ezproxy.utu.fi/10.1177/0969733015584966
- See also: Proposed criteria for reporting the development and evaluation of complex interventions in healthcare (CReDECI): guideline development. — https://doi.org/10.1016/j.ijnurstu.2011.08.003